CLINICAL TRIAL: NCT03994757
Title: Effects of Routines-Based Early Intervention in Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201602004A3
Record Dates: First submitted 2018-12-24; First posted 2019-06-21 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2018-12

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Routine-Based Early Intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRBI group (Experimental)
  Interventions: Behavioral: MRBI
- Control group (Sham Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: MRBI — The activities content is designed according to the children's daily routine and goals. It mainly involves bathing activities, eating activities, dressing activities, game activities, social and communication activities, and according to the needs of parents. In the treatment room, after the therapist and parents discuss the intervention methods and suggestions, they will demonstrate the intervention strategies and methods, and let the parents practice the practice, and the therapist will guide them. After discussing with parents, the therapist will give parents a homework related to children's daily routine, let the parents implement at home, and discuss with parents and record before each intervention.
  Arms: MRBI group
Behavioral: Control — Traditional treatment was directly performed for children in the treatment room by the therapist. The activity content was designed according to the children's goals. After each end of treatment, therapist will give parents a homework related to traditional treatments, let the parents perform at home, and know the parents' performance at home and record before each treatment begins.
  Arms: Control group

SUMMARY:
Autism Spectrum Disorder (ASD) mainly has social and interaction related problems, and repetitive behaviors or interests. In recent years, studies showed that Routine-Based Early Intervention(RBEI) could increase children's development and enhance skills maintenance. Using the International Classification of Functioning, Disability and Health for Children and Youth (ICF-CY) to assess children can identify different factors under systematic analysis, then improving children's physical functions and self-care abilities. Therefore, this study will design RBEI programs for autistic children, and use ICF-CY to assess the efficacy of RBEIin body function, body structure, and participation for children with autism.

DETAILED DESCRIPTION:
Study will enroll 30-40 children with ASD, aged 3-9 years. Children will receive subjective and objective assessment for pre-test, post-test and three-monthfollow-up after treatment. After pre-test, children will be randomized and assigned to either the experimental group or the control group. The experimental group willreceive RBEI and the control group willreceive traditional therapy. The treatment period is 12 weeks, 1-2 times a week, 1-2hours each time, and homework is given during the treatment period, allowing parents to do treatment at home. Post-test will be conducted immediately after the end of treatment period, and homework will continue until three-month follow-up conducts. It is expected that after intervention, the physical function, activities and participation, quality of life of the experimental group will improve and significantly different from the control group.

ELIGIBILITY:
Inclusion Criteria:

* Parents are willing to sign written consent form
* Diagnosed as ASD by doctor
* No neurological disease

Exclusion Criteria:

* Active medical condition
* Progressive or degenerative symptoms or illness

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale(GAS) | baseline, up to 24hours,3-month FU
  It's an individualized assessment tool, setting goals based on the subject's ability and condition, and specifically describe or quantify the progress of the situation, with a view to regularly assessing and understanding whether the subject has progressed or regressed. The scale is a five-point scale from -2 to 2.
Comprehensive Developmental Inventory for Infants and Toddlers(CDIIT) | baseline, up to 24hours,3-month FU
  Applicable to infants and young children aged 3-71 months. It includes the clinical assessment and the parent-report questionnaires. It is used to evaluate the motor, language, cognition, social self-care and other fields of infants and young children. It has good inter-tester reliability, retest reliability, internal consistency, content validity and construction validity. Considering to the comprehensive developmental capacity of children with autism, we assess the overall developmental capacity of children with autism up to nine years oldin this study.

SECONDARY OUTCOMES:
Childhood Asperger Syndrome Test(CAST) | baseline, up to 24hours,3-month FU
  This parent-reported questionnaire is used to screen the autistic characteristic of children with high-function autism or Asperger, including repetitive behavior, social dysfunction and communication deficit, etc. Available age is 4-11. This 2-point questionnaire has 37 items, including 6 non-scoring general developmental items and 31 target items. At the end has additional items identifying whether child has special needs.Retest reliability is .83. Study showed that CAST can screen out 87.5% of children with Asperger.
The Children Autism Rating Scale Second Edition(CARS-2) | baseline, up to 24hours,3-month FU
  This 5-point scale is used to identify whether child is autism. Applicable to preschool children.The internal consistency is .92-.95, inter-rater reliability is .85-.97, and retest reliability is .89-.99.
Clancy Behavior Scale | baseline, up to 24hours,3-month FU
  This 3-point scale is used to screen whether child is autism. Available age is 2-5. The administered time is 10 minutes in average. Total score above 14 shows child has autism tendency and above 23 shows child is autism.It has good sensitivity.
Social Responsiveness Scale(SRS) | baseline, up to 24hours,3-month FU
  Filled out by parents or teachers, the average time is 15-20 minutes. It is used to assess the social barriers of children aged 4-18 and to determine whether a child has autism. It is a four-point scale with a score of 0-3. The internal consistency is 0.91-0.97, retest reliability is 0.84-0.97, inter-rater reliability is 0.76-0.95.
Theory of Mind Inventory-2(ToMI-2) | baseline, up to 24hours,3-month FU
  A questionnaire for assessing children's social cognition ability, which is a five-point questionnaire for continuity. It can be filled out by parents or filled by children with good reading skills and oral skills. Applicable age is 2-13 years old, including 60 topics. Each question is described as a state, including emotional cognition, mental state understanding, pragmatics, etc. The person who fills the mark is marked with a slash on the line of "definitely not"," probably not", "undecided", "probably", and "definitely" to respond. The internal consistency is 0.96.
The Berry-Buktenica Developmental Test of Visual-Motor Integration(VMI) | baseline, up to 24hours,3-month FU
  It is used to assess children's ability to visually recognize and motor coordination. Applicable for 3 years old to adult, and the evaluation time is about 15-20 minutes. It contains high retest reliability and internal consistency.
Preschool Language Impaired Scale(PLS)/ Language Impaired Scale(LS) | baseline, up to 24hours,3-month FU
  It is used to assess whether children have problems in communication, including sound, articulation, intonation, fluency, vocabulary comprehension and expression. Suitable for children from 3 to 5 years old (PLS) and over 5 years old (LS). This 0-1 point measure includes 3 subscales: comprehension, expression and language development. The higher percentile rank represent better outcome. The retest reliability and the inter-tester reliability are 0.91-0.97.
Peabody Picture Vocabulary Test-Revised(PPVT-R) | baseline, up to 24hours,3-month FU
  It is used to assess children's vocabulary comprehension and can also be used as a child intelligence test. Suitable for children from 3-12 years old. The test is based on the number of questions corresponding to the child's physiological age, and the test is tested backward after answering the six questions (the highest level) in the eight consecutive questions, and the test is completed after the eight consecutive questions (basic level). Questions below the basic level are considered correct. Internal consistency and inter-tester reliability are good.
Assessment of preschool children's participation(APCP) / Children Assessment of Participation and Enjoyment andPreferences for Activity of Children(CAPE) | baseline, up to 24hours,3-month FU
  Used to measure children's learning, playing, development skills and personal qualities. Applicable to children aged 2-6 (APCP) and 6-21 (CAPE), the parents score this questionnaire according to the child's performance in the past four months.There are 45 questions in total.First, check if the child have done this activity (1 point means yes, 0 points means no), then check the frequency child doing this activity (1 point, means only once in the last four months, to 7 points, means every day in the past four months). The measurement field includes: 1. Game activities (9 questions) 2. Skill development (15 questions) 3. Sports activities (10 questions) 4. Social activities (11 questions). The measurement aspect includes: diversity, intensity. There is moderate to good internal consistency.
Functional Independence Measure for Children(WeeFIM) | baseline, up to 24hours,3-month FU
  It is used to understand the functional performance of children in the areas of self-care, mobility, and cognition. It is suitable for infants to adolescents. It contains 18 items, involving six functions. The score is from 1 to 7 points, 1 is completely dependent, and 7 is completely independent. Retest reliability and inter-tester reliability are 0.90-0.99.
TNO-AZL Preschool children Quality of Life(TAPQOL)/TNO-AZL Quality of Life Questionnaire(TACQOL) | baseline, up to 24hours,3-month FU
  It is used to assess the health-related quality of life, such as children's motor, communication, emotions, and body structure. Suitable for children from 6 months to 6 years old (TAPQOL) and 6-15 years old (TACQOL). Parents fill in according to the child's condition. First, children or their parents check the frequency of the condition happening (1 ,means never, to 3 , means usually), then check how do children feel when the condition happens (0, means never, to 4 , means not very well).Higher score represent better outcome. Moderate to good retest reliability and inter-tester reliability.
Sensory Profile(SP) | baseline, up to 24hours,3-month FU
  It is used to assess children's sensory processing capabilities, including sensory conditioning, emotional response, sensory processing, etc. Suitable for six-month old child to adults. It is a standardized evaluation tool, which is filled out by the main caregivers. The project score is 1-5 points, the internal consistency reliability is .70-.90, and the inter-tester reliability is .25-.76.
Parenting Stress Index(PSI) | baseline, up to 24hours,3-month FU
  Used to understand parental distress, child distress behaviors and parent-child interaction. Suitable for parents of children under the age of 12. Parents fill in according to subjective feelings and current situation. This 1-5 point measure includes 3 subscales: Parent-Child Dysfunctional Interaction, Difficult Child, and Parent Distress. Higher percentile rank represent worse outcome. Retest reliability and inter-tester reliability is 0.89-0.93.
Swanson, Nolan, and Pelham Questionnaire(SNAP) | baseline, up to 24hours,3-month FU
  It is used to measure the child's inattention, impulsivity or hyperactivity, as well as the status of opposing behavior. Fill in by parents or primary caregivers. This 0-3 point scale includes 26 items. Total scores range from 0 to 78. Higher scores represent a worse outcome. The retest reliability is 0.59-0.72, the internal consistency is 0.88-0.90, and the concurrent validity is 0.56-0.72.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ying Chung, MD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No